CLINICAL TRIAL: NCT07239297
Title: Development and Clinical Application of Deep Learning-Based Retrospective Pathology Foundation Models
Brief Title: Retrospective Pathology Foundation Models
Status: Enrolling by invitation | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-419
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Pancancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Samples Without DNA: Samples retained, with no potential for DNA extraction from any retained samples (e.g., fixed tissue, plasma)

GROUPS / COHORTS (2):
- QFSH external validation dataset: 1000 slides from 1000 eligible individuals were obtained in the Qianfoshan Hospital (QFSH, Jinan, China) between January 2020 and July 2025, which was used to validate the pathology foundation models.
- NFH dataset: We conducted a validation study to compare the diagnostic performance among pathologists, our pathology foundation model, and pathologist-with-AI-assisted diagnosis. This study was initiated at Nanfang Hospital, Southern Medical University (NFHSMU), with patient enrollment from January 1, 2011 to July 31, 2024.

SUMMARY:
By integrating retrospective multimodal data such as pathology and imaging, AI technologies offer novel solutions for disease classification, tumor grading, histological and molecular subtyping, selection of chemotherapy regimens, risk stratification, and treatment-response prediction. This research direction not only deepens our understanding of tumor biological characteristics but also provides essential support for precision medicine and individualized therapy. It holds significant theoretical and practical value and has important implications for mitigating strained medical resources and improving the accuracy of therapeutic decision-making, representing a cutting-edge application with substantial translational potential.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old.
2. Patients with complete pathological slides and clinical information.

Exclusion Criteria:

1.Patients with missing data or specimens not meeting quality control requirements for analysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria comprised patients aged 18-75 years with definitive pathological diagnoses. All cases were retrospectively collected from Nanfang Hospital, Southern Medical University (NFHSMU) .
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Area under ROC curve (AUC) | Diagnostic evaluation will be performed within 1 week when the WSIs are obtained
  Area under the curve

SECONDARY OUTCOMES:
Specificity | Diagnostic evaluation will be performed within 1 week when the WSIs are obtained
  The true negative rate (TNR) of the diagnostic platform, which is the ratio between the number of negative individuals correctly categorized by platform and the total number of actual negative individuals (%).
Sensitivity | Diagnostic evaluation will be performed within 1 week when the WSIs are obtained
  The true positive rate (TPR) of the diagnostic platform, which is the ratio between the number of positive individuals correctly categorized by platform and the total number of actual positive individuals (%).

CONTACTS AND LOCATIONS:
Overall Officials: Li Liang, Study Director — Nanfang Hospital, Southern Medical University
Locations (2):
- China (2):
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Qianfoshan Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No
Requests for the data collected and analyzed in this study will be considered if the application is in line with public benefits and the applicant is willing to sign a data access agreement. Contact can be through the corresponding author.